CLINICAL TRIAL: NCT04876599
Title: IN FOCUS: A Multimodal Mind-Body Intervention for Fear of Recurrence Among Cancer Survivors
Brief Title: Mind-body Resiliency Intervention for Fear of Cancer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Daniel Hall, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-090
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Cancer; Coping Skills; Coping Behavior
Keywords: Cancer; Coping Skills; Coping Behavior
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (IN FOCUS) (Experimental): Participants will be randomly assigned and participate in eight weekly virtual group sessions to learn mind-body, cognitive behavioral, and positive psychology skills.
  Interventions: Behavioral: IN FOCUS
- Usual Care (Active Comparator): Participants will be randomly assigned and receive usual care, which is a referral for virtual group supportive services for cancer survivors provided in the community.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: IN FOCUS — Adapted Resiliency Group Intervention
  Arms: Intervention (IN FOCUS)
Behavioral: Usual Care — Referral to Virtual Group Support
  Arms: Usual Care

SUMMARY:
The purpose of this study is to test the feasibility of a virtual, group mind-body resiliency intervention adapted to target fear of recurrence (FOR) among cancer survivors.

DETAILED DESCRIPTION:
This is a randomized pilot feasibility trial (1:1 intervention versus usual care; a referral to community-based cancer survivor support group) that will use mixed methods (quantitative and qualitative) to evaluate the feasibility, acceptability, and preliminary effects of a virtual, group mind-body resiliency intervention adapted to target fear of recurrence (IN FOCUS) among cancer survivors with clinically elevated fear of recurrence (N = approximately 64).

Patient-reported outcomes on psychological and behavioral outcomes will be measured at T0 (baseline), T1 (post-intervention/approximately two months post-baseline), and T2 (three months post-intervention/approximately five months post-baseline). Exit interviews will be conducted after the T1 survey. Participants are expected to be in the study for approximately five months.

ELIGIBILITY:
Inclusion Criteria:

* History of non-metastatic, localized, or regional solid or blood malignancy(ies)
* Completion of primary cancer treatment (i.e., radiation, surgery, chemotherapy) and/or current use of long-term maintenance hormonal or biologic therapy
* Age ≥18 years
* Elevated fear of recurrence (FCRI severity score ≥16)
* MGB/BIDMC Medical Record Number (MRN)

Exclusion Criteria:

* Self-reported inability to speak and write in English
* Undertreated serious mental illness as defined by history of suicidality, psychosis, and/or psychiatric hospitalization in the past year
* Inability to access technology and/or sufficient internet to participate virtual groups sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hall, PhD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Massachusett General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mass General at Emerson Hospital -- Bethke, Concord, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Daniel L. Hall, PhD (hall@mgh.harvard.edu). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Christie AJ, Bolden C, Park ER, Yeh GY, O'Cleirigh C, Peppercorn J, Denninger JW, Hirschberg AM, Lee H, Markwart M, Siefring E, Mizrach HR, Bullock AJ, Hall DL. Managing, not lessening, uncertainty: a novel mind-body intervention for fear of cancer recurrence. J Cancer Surviv. 2025 Sep 1. doi: 10.1007/s11764-025-01886-2. Online ahead of print. PMID 40887510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (IN FOCUS) | Usual Care
Started | 32 | 32
Follow up Survey #1 | 31 | 31
Exit Interview | 29 | 30
Follow up Survey #2 | 29 | 29
Completed | 28 (Within the IN FOCUS arm, one participant missed the deadline to complete the T1 survey, two participants declined the exit interview and T2 survey (time constraints), and an additional participant missed the exit interview and T2 survey.) | 29 (Within the Usual Care Control arm, one participant declined study participation (dissatisfaction with randomization), one participant declined the exit interview and T2 survey (time constraints), and one participant declined the T2 survey.)
Not Completed | 4 | 3
Not completed — Missed | 2 | 0
Not completed — Declined | 2 | 3

BASELINE CHARACTERISTICS:
Population: All participants who consented and completed the baseline survey
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (IN FOCUS) | Usual Care | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (14.7) | 53.7 (12.7) | 52.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could be included in more than one Race/Ethnicity category/row.
  Participants
    Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Black or African American | 4 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    White | 29 | 30 | 59
    Other | 2 | 1 | 3
    Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Retention Rate
Description: The primary metric for assessing feasibility will be retention at the initial follow-up assessment (≥70% survey completion). For descriptive purposes, secondary exploratory metrics of feasibility will include reasons for ineligibility, refusal, or dropping out will be measured, as will rates of enrollment, ratio of screened-to-eligible, attendance (e.g., ≥75% of intervention sessions attended), self-reported adherence to relaxation skills practice, and interventionist fidelity. Exit interviews will use open-ended questions to assess the feasibility of attending virtual sessions.
Time Frame: Baseline to approximately 2 months
Measure: Count of Participants; unit: Participants
Groups:
- IN FOCUS: Participants will be randomly assigned and participate in eight weekly virtual group sessions to learn mind-body, cognitive behavioral, and positive psychology skills.
  IN FOCUS: Adapted Resiliency Group Intervention
Arm/Group | IN FOCUS | Usual Care
Number analyzed (Participants) | 32 | 32
Participants | 31 | 31

2. Primary Outcome: Acceptability: 5 Item Measure of Enjoyableness, Convenience, Helpfulness, Odds of Future Use, and Overall Satisfaction
Description: As a primary quantitative acceptability outcome, participants will be asked to rate the enjoyableness, convenience, helpfulness, odds of future use, and overall satisfaction (1=very low to 5=very high) of the intervention.
Time Frame: Baseline to approximately 2 months
Population: This acceptability metric was assessed within the intervention arm only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Acceptability Items: IN FOCUS participants who responded to the acceptability measure.
Arm/Group | Acceptability Items
Number analyzed (Participants) | 30
score on a scale
  Enjoyableness | 4.33 (.71)
  Convenience | 4.57 (.82)
  Helpfulness | 4.00 (1.02)
  Odds of Future Skills Use | 4.33 (1.03)
  Overall Satisfaction | 4.20 (.92)

3. Secondary Outcome: Fear of Cancer Recurrence
Description: Fear of cancer recurrence (FCR) severity will be measured using the 9-item Fear of Cancer Recurrence Inventory severity subscale. Scores range from 0-36 with higher scores indicating greater FCR severity. To supplement this measure, open-ended questions in the exit interview will assess perceived changes in FCR.
Time Frame: Baseline, approximately 2 months, approximately 5 months
Population: Not all surveys were returned.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN FOCUS | Usual Care
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 23.62 (4.19) | 22.22 (4.88)
  2 Months: number analyzed (Participants) | 31 | 31
  2 Months | 19.74 (4.54) | 20.90 (5.34)
  5 Months: number analyzed (Participants) | 29 | 29
  5 Months | 20.66 (5.21) | 19.27 (6.08)

4. Secondary Outcome: Resiliency
Description: Resiliency will be measured using the 23-item Current Experiences Scale. Subscale scores and total scores (range from 0-115) will be computed, with higher scores indicating higher resiliency.
Time Frame: Baseline, approximately 2 months, approximately 5 months
Population: Not all surveys were returned.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN FOCUS | Usual Care
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 71.05 (14.00) | 75.23 (14.05)
  2 Months: number analyzed (Participants) | 29 | 31
  2 Months | 76.24 (11.89) | 76.80 (15.51)
  5 Months: number analyzed (Participants) | 28 | 29
  5 Months | 81.05 (11.66) | 75.45 (16.34)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from all participants (n=64) and monitored throughout the duration of their study participation, approximately 5 months.
Arm/Group | Intervention (IN FOCUS) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04876599/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04876599/SAP_001.pdf